CLINICAL TRIAL: NCT04775524
Title: An Arts-based Intervention With Healthcare Workers: Storytelling Through Music to Address Work Related Emotions (AWARENESS Trial)
Brief Title: AWARENESS Trial (AWARENESS) of Storytelling Through Music in Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Carolyn Phillips, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-710
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Stress; Post Traumatic Stress Disorder; Work Related Stress
Keywords: Stress; Post Traumatic Stress Disorder; Work Related Stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Occupational Stress | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Storytelling Through Music (STM) (Experimental): Participants will be randomized into two (2) groups: Storytelling Through Music (STM) and Waitlist (Storytelling Through Music-Hybrid)
  Storytelling Through Music (STM) group will participate in the study for a total of 19 weeks with 6 weeks of the STM program and 3 months follow up.
  * Storytelling Through Music (STM) utilizes multiple modalities including storytelling, reflective writing, self-care skills (i.e., breathing exercises, meditation, self-compassion, body scans), and songwriting.
    * Weeks 1-4: participants are led through weekly writing workshop over an online platform (i.e., Zoom or an equivalent) to develop their stories. Simultaneous with the writing sessions are 10-minute self-care lessons
    * Week 5: Participants will be paired with a professional songwriter who will put their story into a song.
    * Week 6: During the last week, participants will have one more writing workshop to debrief about the intervention.
  Interventions: Behavioral: Storytelling Through Music (STM)
- Wait List / Storytelling Through Music-Hybrid (Experimental): Participants will be randomized into two (2) groups: Storytelling Through Music (STM) and Waitlist (Storytelling Through Music-Hybrid)
  Waitlist control group (Storytelling Through Music-Hybrid) will participate in the study for a total of 13 weeks with 2 weeks of Storytelling Through Music-Hybrid program and 11 weeks of follow up .
  * Storytelling Through Music-Hybrid involves participants listening to songs created for other healthcare professionals for 2 weeks.
  Interventions: Behavioral: Wait List / Storytelling Through Music-Hybrid

INTERVENTIONS:
Behavioral: Storytelling Through Music (STM) — 6 week expressive arts-based program
  Arms: Storytelling Through Music (STM)
Behavioral: Wait List / Storytelling Through Music-Hybrid — 2 week song listening program
  Arms: Wait List / Storytelling Through Music-Hybrid

SUMMARY:
This research study is examining the feasibility and effectiveness of an online version of the Storytelling Through Music (STM) program with oncology nurses who have worked during the COVID-19 pandemic.

DETAILED DESCRIPTION:
This study employs a two-group, randomized controlled trial design that will utilize quantitative and qualitative methods to evaluate the feasibility and intervention effect of an alternative delivery (online) of the Storytelling Through Music program (STM).

Previous study of In-person delivery of Storytelling Through Music program STM with oncology nurses found it to be feasible and beneficial to coping with stress and work-related emotions.

The research study procedures include: screening for eligibility and study intervention including follow-up surveys.

Participants will be randomized into two (2) groups: Storytelling Through Music (STM) and Waitlist (Storytelling Through Music-Hybrid)

STM group: Participants are led through a writing workshop over an online platform (i.e., Zoom or an equivalent) to develop their story. Simultaneous with the writing sessions are 10-minute self-care lessons. At the end of the development workshop, each participant will be paired with a songwriter who will turn participant stories into songs. A final workshop will be held for participants to debrief about the emotional experience of participating in the Storytelling Through Music program (STM)

Waitlist control group (Storytelling Through Music-Hybrid), will listen to songs created by healthcare workers in the Storytelling Through Music program (STM) for 2 weeks.

Participation length will be based on the randomized group assignment, a total of 19 weeks for the STM group and 13 weeks for the waitlist group.

It is expected that about 50 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study is as follows: a) >18 years old; b) licensed oncology nurse; c) provided direct patient care during COVID-19 pandemic.

Exclusion Criteria:

* Key exclusion criteria include: a) have previously participated in the STM intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | 6 weeks
  Primary endpoint is feasibility using visual analog scale Descriptive statistics will be used on the visual analog scale questions for analysis of feasibility. This intervention will be deemed feasible if 85% of the intervention is completed and 60% find it acceptable.
Acceptability of intervention | 6 weeks
  Additional primary endpoint is acceptability using descriptive qualitative data.
  Open-ended questions will prompt participants to provide insights into quantitative findings and the acceptability of the intervention.
  This intervention will be deemed feasible if 85% of the intervention is completed and 60% find it acceptable.

SECONDARY OUTCOMES:
Self-awareness | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  Self-Reflection and Insight Scale; range is 12-72; higher score means better outcome.
Post-traumatic stress | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  Impact of Event Scale-Revised; range is 0-88; lower score is better outcome.
Self-compassion | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  Self-Compassion Scale; range is 26-130; higher score is better outcome.
Anxiety | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  PROMIS Anxiety Scale (Short-form 6); range is 5-30; lower score is better outcome.
Depression | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  PROMIS Depression Scale (Short-form 8); range is 8-40; lower score is better outcome.
Insomnia | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  Insomnia Severity Index; range is 0-28; lower score is better outcome
Loneliness | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  UCLA Loneliness Scale; range is 0-60; lower score is better outcome.
Post-traumatic growth | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  Post-Traumatic Growth Index; range is 0-105; lower score is better outcome.
Professional Quality of Life | 6 weeks (both groups), 11 weeks (both groups), 19weeks (intervention group only)
  Professional Quality of Life Scale; 3 separate subscale scores=burnout (range is 10-50; lower score equals better outcome); Secondary traumatic stress (range is 10-50; lower score equals better outcome); Compassion satisfaction (range is 10-50; higher score equals better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Phillips, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Phillips CS, Morris SE, Woods H, Mazzola E, Xiong N, Young C, Stuifbergen A, Hammer M, Ligibel J. A Randomized Controlled Feasibility Study to Evaluate the Online Delivery of Storytelling Through Music With Oncology Nurses. Cancer Nurs. 2024 Dec 19. doi: 10.1097/NCC.0000000000001441. Online ahead of print. PMID 39701577